CLINICAL TRIAL: NCT05965908
Title: Effect of Liraglutide on Different Parameters (Clinical , Metabolic and Hormonal) in Obese Women With Polycystic Ovary Syndrome
Brief Title: Effect of Liraglutide in Obese Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Liraglutide Polycystic Ovary
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Polycystic Ovary
Keywords: polycystic ovary; liraglutide
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Liraglutide; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- liraglutide (Experimental): Saxenda® starting dose is 0.6 mg per day for 1 week.1. Patients increase the dose by 0.6 mg each week until the full maintenance dose of 3 mg is reached
  Interventions: Drug: liraglutide
- metformin (Active Comparator): the patient is given Glucophage 1000 mg tab once daily after lunch for 1month
  Interventions: Drug: Metformin
- control (No Intervention): not given any drug

INTERVENTIONS:
Drug: liraglutide — glucagon-like peptide 1 receptor agonist
  Other Names: saxenda ampoules
  Arms: liraglutide
Drug: Metformin — biguanide antihyperglycemic
  Other Names: Glucophage 1000mg
  Arms: metformin

SUMMARY:
The aim of this study is to compare the hormonal, metabolic and clinical effects of metformin and liraglutide in infertile women with PCOs.

DETAILED DESCRIPTION:
It is a Prospective randomized controlled trial .The study will include 80 randomly selected infertile women aged between 18 and 45 years, from Gynecology and obstetrics department Beni-Suef University Hospital whom diagnosed with polycystic ovarian syndrome (PCOS), The study will include two groups; each group consists of 40 patients:-

* Group1 (n=40) will be treated by liraglutide monotherapy.
* Group 2 (n=40) will be treated by metformin monotherapy.
* Group 3 (n=40) will be a control group.

To assess the metabolic effect of each treatment, the following parameters will be assessed before and after the treatment

* To assess the hormonal effect of each treatment, the following tests will be assessed before and after treatment
* Total Testosterone (TT)
* Dehydroepiandrosterone (DHEA)

To assess the clinical effect of the drugs, the following will be assessed before and after treatment:

The number of medium size follicles and large size follicles and the endometrium thickness were assessed on the tenth or eleventh day of menstruation. The chemical and clinical pregnancy rates were evaluated

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 45 years
* PCO

Exclusion Criteria:

1. congenital adrenal hyperplasia
2. poorly controlled thyroid disease
3. Taking antidiabetic drugs which can affect insulin resistance
4. chronic kidney disease and history of recurrent urinary tract infections
5. liver dysfunction
6. documented use of oral hormonal contraceptives and hormone-releasing implants

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Body weight loss | 1 months
  basal body weight - body weight reached after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Study Director — Clinical Pharmacy Faculty of Pharmacy Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected data
Supporting Information: Study Protocol, SAP